CLINICAL TRIAL: NCT05309018
Title: Implantation of an Advanced Practice Nurse in the Complex Care Pathway of Patients Followed for AML Treated With Oral Targeted Therapy
Brief Title: Implantation of an Advanced Practice Nurse in the Complex Care Pathway of Patients With AML
Acronym: LAMIPA
Status: Withdrawn | Type: Observational
Why Stopped: investigator's unavailability
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-07Obs-CHRMT
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Myeloid Leukemia
Keywords: Advanced Practice Nurse; Acute Myeloid Leukemia,
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Interviews
- medical staff
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Semi-structured interview about perceptions and expectations of APN participation in AML monitoring according to patient and to care team.

SUMMARY:
Advanced Practice Nurse (APN) is a new contributor in the French healthcare system. APN is part of a multidisciplinary team and aim to monitor patients under the coordination of the doctor particularly in onco-hematology. The aim of the study is to describe the different perceptions and expectations of APN monitoring according to patients with acute myeloid leukemia (AML) and their care team.

This study will involve 10 patients, recruited over a provisional period of 5 months and 25 member of care team. Patients and their care team will be asked about their perceptions and expectations of APN participation in (AML monitoring) during a semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patient with AML
* Treated with a new targeted oral therapy as monotherapy or in combination:

  * Venetoclax* in combination with ivosidenib (IDH1 inhibitor)
  * Onureg* (azacitin: pyrimidine analogue)
  * Venetoclax (BCL-2 protein inhibitor) in combination with subcutaneous azacitin
* Whose follow-up is provided alternately by a hematologist and an IPA.
* Affiliated to a social security scheme

Exclusion Criteria:

* Moderate or severe cognitive impairment
* Language barrier
* Other communication disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with MLA Care team
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Perception of patient | Within 1 month
  Semi-structured interview about perceptions and expectations of Advanced Practice Nurse (APN) participation in acute myeloid leukemia (AML) monitoring according to patient.

SECONDARY OUTCOMES:
Perception of care team | Within 1 month
  Semi-structured interview about perceptions and expectations of Advanced Practice Nurse (APN) participation in acute myeloid leukemia (AML) monitoring according to care team.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer HUET, Principal Investigator — CHR Metz Thionville Hopital de Mercy